CLINICAL TRIAL: NCT02220556
Title: Evaluation of Different Analysis Methods for Circulating Tumor Cells, Circulating Endothelial Cell, and Circulating Tumor DNA in Patient Followed for a Tumoral Pathology
Acronym: CTC-CEC-ADN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IC 2010-01
Record Dates: First submitted 2014-08-08; First posted 2014-08-20 (Estimated); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Solid Tumor, Adult
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Blood sampling

SUMMARY:
Fifteen cohorts will be opened. Each cohort will explore one analysis method and/or tumoral type. Up to 50 patient can be included into each cohort.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or more
* Performance status from 0 to 4
* Patient treated followed for histologically confirmed solid tumor type of any of these localization : breast, prostate, uterus, ovary, colon, lung, head and neck, melanoma.
* Informed consent form signed.

Exclusion Criteria:

* Patient with history of other invasive cancer within 5 years.
* Patient treated for any non-invasive cancer
* Patient individually deprived of liberty or placed under the authority of a tutor
* Geographical condition potentially preventing compliance with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2010-12; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
CTC, CEC or ctDNA incidence | 3 years
  number of CTC or CEC in 7.5ml of blood

SECONDARY OUTCOMES:
CTC and CEC molecular characterization | 3 years
  This outcome is self-explanatory.
Circulating tumor DNA (ctDNA) detection and quantification | 3 years
  plasma mutation detection (number of copy)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Yves Pierga, Prof., Principal Investigator — Institut Curie; François-Clément Bidard, MD, PhD, Study Chair — Institut Curie
Locations (3):
- France (3):
  - Institut Curie, Paris
  - Institut Mutualiste Montsouris, Paris
  - Institut Curie, Saint-Cloud

REFERENCES:
- [Background] Cabel L, Jeannot E, Bieche I, Vacher S, Callens C, Bazire L, Morel A, Bernard-Tessier A, Chemlali W, Schnitzler A, Lievre A, Otz J, Minsat M, Vincent-Salomon A, Pierga JY, Buecher B, Mariani P, Proudhon C, Bidard FC, Cacheux W. Prognostic Impact of Residual HPV ctDNA Detection after Chemoradiotherapy for Anal Squamous Cell Carcinoma. Clin Cancer Res. 2018 Nov 15;24(22):5767-5771. doi: 10.1158/1078-0432.CCR-18-0922. Epub 2018 Jul 27. PMID 30054279
- [Background] Cabel L, Decraene C, Bieche I, Pierga JY, Bennamoun M, Fuks D, Ferraz JM, Lefevre M, Baulande S, Bernard V, Vacher S, Mariani P, Proudhon C, Bidard FC, Louvet C. Limited Sensitivity of Circulating Tumor DNA Detection by Droplet Digital PCR in Non-Metastatic Operable Gastric Cancer Patients. Cancers (Basel). 2019 Mar 21;11(3):396. doi: 10.3390/cancers11030396. PMID 30901876